CLINICAL TRIAL: NCT04260399
Title: AROMA Study: Anxiety Reduction During Office Procedural Medicine Using Aromatherapy
Brief Title: Anxiety Reduction During Office Procedural Medicine Using Aromatherapy
Acronym: AROMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Thythy Pham, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 213113
Record Dates: First submitted 2020-01-27; First posted 2020-02-07 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Anxiety; Anxiety State; Procedural Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Patients are randomized to lavender aromatherapy or saline placebo aromatherapy using a 1:1 random block allocation
Masking Description: This trial is not blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lavender Aromatherapy (Experimental): Passive exposure via an ambient essential oil diffuser to lavender aromatherapy
  Interventions: Other: Lavender Aromatherapy
- Placebo Aromatherapy (Placebo Comparator): Passive exposure via an ambient essential oil diffuser to saline water aromatherapy
  Interventions: Other: Placebo Aromatherapy

INTERVENTIONS:
Other: Lavender Aromatherapy — Participants in the experimental group will be passively exposed to lavender essential oil
  Arms: Lavender Aromatherapy
Other: Placebo Aromatherapy — Participants in the control group will be passively exposed to saline water aromatherapy
  Arms: Placebo Aromatherapy

SUMMARY:
This goal of this study is to assess whether lavender aromatherapy during gynecologic and urogynecologic outpatient procedures is associated with a decrease in patient anxiety levels. Based on similar interventions in other specialties of medicine, the investigators hypothesize that patients exposed to lavender aromatherapy during their procedure will have less anxiety than those who are not exposed to lavender aromatherapy.

DETAILED DESCRIPTION:
Patients who present to the Loyola Urogynecology office for an outpatient procedure will be invited to participate. Patients who consent to participate will be asked to complete pre-procedure questionnaires including an assessment of their level of procedural anxiety. Subsequently, patients will be randomized to receive either lavender aromatherapy or saline aromatherapy (placebo) during their procedure. Post-procedural levels of anxiety will then be assessed. Changes between pre- and post-procedural anxiety will be compared between the treatment and placebo control groups.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing the following gynecologic/urogynecologic office procedures: colposcopy, loop electrical excision procedure (LEEP), endometrial biopsy, intrauterine device (IUD) insertion, hysteroscopy, Nexplanon removal, cystoscopy, urodynamics, botox intravesical injection, and transurethral bulking injection
* English speaking
* Ability to complete questionnaires

Exclusion Criteria:

* Pregnancy
* Allergy to lavender scent
* Lung disease including asthma or chronic lung disease
* Anosmia or problems related to smell
* Chronic headaches or migraines
* Inability to complete questionnaires

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Change in state trait anxiety level | Immediate post-procedure
  Participants' change in state anxiety from pre-procedure to post-procedure will be measured using the State-Trait Anxiety Inventory (STAI-Y1). The STAI-Y1 is a 20 item questionnaire that asks participants to rate their state anxiety. The scale ranges from 20 to 80 points with higher scores indicating worse anxiety. The change score is calculated by subtracting the pre-procedure STAY-YI score from the post-procedure STAY-YI score to create a delta STAI-Y1 score.

CONTACTS AND LOCATIONS:
Overall Officials: Thythy Pham, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Bailey L. Strategies for decreasing patient anxiety in the perioperative setting. AORN J. 2010 Oct;92(4):445-57; quiz 458-60. doi: 10.1016/j.aorn.2010.04.017. PMID 20888947
- [Background] Hilden M, Sidenius K, Langhoff-Roos J, Wijma B, Schei B. Women's experiences of the gynecologic examination: factors associated with discomfort. Acta Obstet Gynecol Scand. 2003 Nov;82(11):1030-6. doi: 10.1034/j.1600-0412.2003.00253.x. PMID 14616277
- [Background] Handelzalts JE, Krissi H, Levy S, Broitman M, Binyamin L, Peled Y. Multidimensional associations of pain and anxiety before and after colposcopy. Int J Gynaecol Obstet. 2015 Dec;131(3):297-300. doi: 10.1016/j.ijgo.2015.05.038. Epub 2015 Sep 6. PMID 26386494
- [Background] Seklehner S, Engelhardt PF, Remzi M, Fajkovic H, Saratlija-Novakovic Z, Skopek M, Resch I, Duvnjak M, Hruby S, Wehrberger C, Librenjak D, Hubner W, Breinl E, Riedl C. Anxiety and depression analyses of patients undergoing diagnostic cystoscopy. Qual Life Res. 2016 Sep;25(9):2307-14. doi: 10.1007/s11136-016-1264-z. Epub 2016 Mar 17. PMID 26984467
- [Background] Biardeau X, Lam O, Ba V, Campeau L, Corcos J. Prospective evaluation of anxiety, pain, and embarrassment associated with cystoscopy and urodynamic testing in clinical practice. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):104-110. doi: 10.5489/cuaj.4127. PMID 28515809
- [Background] Garcia-Perdomo HA, Montealegre Cardona LM, Cordoba-Wagner MJ, Zapata-Copete JA. Music to reduce pain and anxiety in cystoscopy: a systematic review and meta-analysis. J Complement Integr Med. 2018 Oct 12;16(3):/j/jcim.2019.16.issue-3/jcim-2018-0095/jcim-2018-0095.xml. doi: 10.1515/jcim-2018-0095. PMID 30312164
- [Background] Kim JW, Kim HJ, Park YJ, Kang SG, Park JY, Bae JH, Kang SH, Park HS, Moon DG, Cheon J, Lee JG, Kim JJ, Oh MM. The effects of a heating pad on anxiety, pain, and distress during urodynamic study in the female patients with stress urinary incontinence. Neurourol Urodyn. 2018 Mar;37(3):997-1001. doi: 10.1002/nau.23326. Epub 2018 Mar 8. PMID 29516595
- [Background] Kwon WA, Lee JW, Seo HK, Oh TH, Park SC, Jeong HJ, Seo IY. Hand-Holding during Cystoscopy Decreases Patient Anxiety, Pain, and Dissatisfaction: A Pilot Randomized Controlled Trial. Urol Int. 2018;100(2):222-227. doi: 10.1159/000485745. Epub 2017 Dec 22. PMID 29275402
- [Background] Kim JT, Ren CJ, Fielding GA, Pitti A, Kasumi T, Wajda M, Lebovits A, Bekker A. Treatment with lavender aromatherapy in the post-anesthesia care unit reduces opioid requirements of morbidly obese patients undergoing laparoscopic adjustable gastric banding. Obes Surg. 2007 Jul;17(7):920-5. doi: 10.1007/s11695-007-9170-7. PMID 17894152
- [Background] Kim JT, Wajda M, Cuff G, Serota D, Schlame M, Axelrod DM, Guth AA, Bekker AY. Evaluation of aromatherapy in treating postoperative pain: pilot study. Pain Pract. 2006 Dec;6(4):273-7. doi: 10.1111/j.1533-2500.2006.00095.x. PMID 17129308
- [Background] Perry R, Terry R, Watson LK, Ernst E. Is lavender an anxiolytic drug? A systematic review of randomised clinical trials. Phytomedicine. 2012 Jun 15;19(8-9):825-35. doi: 10.1016/j.phymed.2012.02.013. Epub 2012 Mar 29. PMID 22464012
- [Background] Kang HJ, Nam ES, Lee Y, Kim M. How Strong is the Evidence for the Anxiolytic Efficacy of Lavender?: Systematic Review and Meta-analysis of Randomized Controlled Trials. Asian Nurs Res (Korean Soc Nurs Sci). 2019 Dec;13(5):295-305. doi: 10.1016/j.anr.2019.11.003. Epub 2019 Nov 16. PMID 31743795
- [Background] Trambert R, Kowalski MO, Wu B, Mehta N, Friedman P. A Randomized Controlled Trial Provides Evidence to Support Aromatherapy to Minimize Anxiety in Women Undergoing Breast Biopsy. Worldviews Evid Based Nurs. 2017 Oct;14(5):394-402. doi: 10.1111/wvn.12229. Epub 2017 Apr 10. PMID 28395396
- [Background] Franco L, Blanck TJ, Dugan K, Kline R, Shanmugam G, Galotti A, von Bergen Granell A, Wajda M. Both lavender fleur oil and unscented oil aromatherapy reduce preoperative anxiety in breast surgery patients: a randomized trial. J Clin Anesth. 2016 Sep;33:243-9. doi: 10.1016/j.jclinane.2016.02.032. Epub 2016 May 5. PMID 27555173
- [Background] Karaman T, Karaman S, Dogru S, Tapar H, Sahin A, Suren M, Arici S, Kaya Z. Evaluating the efficacy of lavender aromatherapy on peripheral venous cannulation pain and anxiety: A prospective, randomized study. Complement Ther Clin Pract. 2016 May;23:64-8. doi: 10.1016/j.ctcp.2016.03.008. Epub 2016 Mar 25. PMID 27157961
- [Background] Hu PH, Peng YC, Lin YT, Chang CS, Ou MC. Aromatherapy for reducing colonoscopy related procedural anxiety and physiological parameters: a randomized controlled study. Hepatogastroenterology. 2010 Sep-Oct;57(102-103):1082-6. PMID 21410035
- [Background] Muzzarelli L, Force M, Sebold M. Aromatherapy and reducing preprocedural anxiety: A controlled prospective study. Gastroenterol Nurs. 2006 Nov-Dec;29(6):466-71. doi: 10.1097/00001610-200611000-00005. PMID 17273013
- [Background] S PK, Aafaque S, S S, N N. Effect of Aromatherapy on Dental Anxiety Among Orthodontic Patients: A Randomized Controlled Trial. Cureus. 2019 Aug 2;11(8):e5306. doi: 10.7759/cureus.5306. PMID 31592362
- [Background] Tugut N, Demirel G, Baser M, Ata EE, Karakus S. Effects of lavender scent on patients' anxiety and pain levels during gynecological examination. Complement Ther Clin Pract. 2017 Aug;28:65-69. doi: 10.1016/j.ctcp.2017.05.006. Epub 2017 May 13. No abstract available. PMID 28779939